CLINICAL TRIAL: NCT03920761
Title: Evaluation of Technologies for Neonates in Africa
Acronym: ETNA
Status: Completed | Type: Observational
Sponsor: Save the Children (Other)
Collaborators: Aga Khan University (Other); University of British Columbia (Other); EarlySense Ltd. (Industry); SWICA (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ETNA
Record Dates: First submitted 2019-04-03; First posted 2019-04-19 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Neonatal Physiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: EarlySense Insight system — a small piezoelectric sensor pad that can be placed under the mattress and provide contact-free monitoring by measuring and recording a patient's vital signs and motion parameters
Device: Advanced Neonatal Epidermal System — a system of neonatal non-invasive adhesive sensors. Sensors are attached directly on the patient's body and are capable of continuously measuring and recording heart rate, respiratory rate, oxygen saturation, and skin temperature.

SUMMARY:
This is a diagnostic accuracy evaluation and clinical feasibility study of investigational devices (EarlySense and ANNE systems) in a neonatal high dependency unit (nHDU) in a private teaching hospital and a government maternity hospital in Nairobi, Kenya. Neonates who are admitted for routine observation and care will be enrolled.

DETAILED DESCRIPTION:
To further reduce neonatal mortality rate in low resource settings (LRS) in Africa, research is needed to develop and optimize innovations in neonatal care, specifically technologies that are low cost, operator-independent, and highly efficient. The purpose of this study is to produce information and data regarding the performance of two existing multiparameter continuous physiological monitoring devices developed by device developers, EarlySense and Sonica. The clinical trial is intended to provide evidence to establish whether these investigational devices can reliably and accurately measure vital signs in neonates (when compared to verified reference devices) and to assess the feasibility, usability and acceptability of these devices for use in neonates in a LRS in Africa.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female neonate, corrected age of ≤ 28 days.
2. Willingness and ability of neonate's caregiver to provide informed consent and to be available for follow-up for the planned duration of the study.

Exclusion Criteria:

1. Receiving mechanical ventilation or continuous positive airway pressure (CPAP).
2. Skin abnormalities in the nasopharynx and/or oropharynx.
3. Contraindication to application of skin sensors.
4. Known arrhythmia.
5. Presence of a congenital abnormality requiring major surgical intervention.
6. Any medical or psychosocial condition or circumstance that, in the opinion of the investigators, would interfere with the conduct of the study or for which study participation might jeopardize the neonate's health.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates enrolled in the study will be representative of the ethnic demographics in Nairobi, Kenya. Both female and male neonates will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 575 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Determine the accuracy the investigational devices: Agreement of the relevant measurement | Measurements will be collected at one minute intervals for a minimum of 1 hour
  Agreement of the relevant measurement parameters of interest between the investigational device and the reference device(s) at each observation
Determine the clinical feasibility of the investigational devices: Agreement of clinical event detection | Measurements collected at one minute intervals for a minimum of 1 hour
  Agreement of clinical event detection between the investigational device and the reference device(s) at each observation.
Assess the feasibility, usability and acceptability of the investigational device: questionnaire | One 30 minute in-depth interview
  Qualitative questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ansermino, Principal Investigator — BC Children's Hospital, Canada
Locations (2):
- Kenya (2):
  - Aga Khan University Hospital, Nairobi, Nairobi
  - Pumwani Maternity Hospital, Nairobi

IPD SHARING:
Plan to Share IPD: Undecided
If in the future data sharing is needed, the study will establish appropriate data transfer agreements with other researchers and only de-identified data will be shared.

REFERENCES:
- [Derived] Kinshella MW, Naanyu V, Chomba D, Waiyego M, Rigg J, Coleman J, Hwang B, Ansermino JM, Macharia WM, Ginsburg AS. Qualitative study exploring the feasibility, usability and acceptability of neonatal continuous monitoring technologies at a public tertiary hospital in Nairobi, Kenya. BMJ Open. 2022 Jan 11;12(1):e053486. doi: 10.1136/bmjopen-2021-053486. PMID 35017248
- [Derived] Wang D, Macharia WM, Ochieng R, Chomba D, Hadida YS, Karasik R, Dunsmuir D, Coleman J, Zhou G, Ginsburg AS, Ansermino JM. Evaluation of a contactless neonatal physiological monitor in Nairobi, Kenya. Arch Dis Child. 2022 Jun;107(6):558-564. doi: 10.1136/archdischild-2021-322344. Epub 2021 Nov 5. PMID 34740876
- [Derived] Ginsburg AS, Nkwopara E, Macharia W, Ochieng R, Waiyego M, Zhou G, Karasik R, Xu S, Ansermino JM. Evaluation of non-invasive continuous physiological monitoring devices for neonates in Nairobi, Kenya: a research protocol. BMJ Open. 2020 Apr 12;10(4):e035184. doi: 10.1136/bmjopen-2019-035184. PMID 32284391